CLINICAL TRIAL: NCT01125449
Title: Phase 2 Study of High Dose Ascorbic Acid in Solid Tumor Disease
Brief Title: Study of High Dose Intravenous (IV) Ascorbic Acid in Measurable Solid Tumor Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Awaiting response from FDA as to status of parenteral ascorbic acid manufactured by Bioniche (Ireland).
Sponsor: Situs Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L500HD
Record Dates: First submitted 2010-05-16; First posted 2010-05-18 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma; Adenocarcinoma; Carcinoma; Multiple Myeloma; Desmoplastic Small Round Cell Tumor
Keywords: ascorbic acid; vitamin C; antioxidants; vitamins
MeSH Terms: conditions — Sarcoma; Adenocarcinoma; Carcinoma; Multiple Myeloma; Desmoplastic Small Round Cell Tumor | interventions — Ascorbic Acid; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous IVC Intervention (Other): Intravenous ascorbic acid, 1.5g/kg at an infusion rate not to exceed 250mg/min.
  Interventions: Drug: Ascorbic acid (vitamin C)

INTERVENTIONS:
Drug: Ascorbic acid (vitamin C) — Intravenous administration of up to 1.5gm/kg of ascorbic acid, twice weekly for up to 12-weeks.
  Other Names: Bioniche ascorbic acid, parenteral, 500mg/ml

SUMMARY:
The study is designed to determine if high doses of intravenous ascorbic acid (vitamin C) can be effective in managing solid tumor diseases. Secondary goals are determination of any palliative effects and improvement of quality of life of patients.

DETAILED DESCRIPTION:
Ascorbic acid has demonstrated selective cytotoxicity in cancer cells in vitro, while sparing normal cells from its peroxidative effects. This study will examine the effect, if any, of the drug when dosed in patients at a level sufficient to achieve transient serum states of 400mg/dl. Safety of the drug has been shown in a Phase I study when dosed as high as 1.5gm/kg. Patients will be treated twice weekly for 12 weeks (24-cycles) and evaluated for response using RECIST criteria. Patients showing stable disease or objective response will remain on study for up to one year or until absence of measurable disease or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at time of entry on study
* Disease extent confirmed and documented by CT scan within 45 days of entry on study
* normal glucose 6-phosphate dehydrogenase
* no current calcium oxalate nephrolithiasis with the potential to reduce urinary flow
* ability to understand the informed consent process and to give informed consent to treatment
* measurable solid tumor neoplastic disease (using RECIST criteria)
* life expectancy greater than 8-weeks
* will agree to undergo central line placement (examples are: port-a-catheter, central venous catheter, percutaneously inserted central catheter [PICC] line placement). Patient or regular caregiver must be able to maintain flush central line as directed by study physician. (Study center will provide periodic site dressing changes as required)
* Failed curative therapy or patient ineligible for definitive curative therapy
* Karnofsky performance status of at least 40

Exclusion Criteria:

* any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, or ECG at baseline which, in the opinion of the investigator, may put the subject at risk because of his/her participation in the study
* use of any nicotine product including nicotine patches/gum
* unstable angina not well managed with medication
* history of calcium oxalate stone formation
* pregnancy or nursing of an infant
* any psychiatric disorder by history or examination that would prevent completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment | 12-weeks
  Survival as a result of efficacy of treatment will be evaluated at 12-weeks. Efficacy is evaluated using RECIST criteria to determine disease response by PET/CT scan interpretation, lab studies and current good clinical practice methodologies for solid tumor interventional treatment.

SECONDARY OUTCOMES:
Patient self-assessment of Quality of Life at 12-weeks | 12-weeks
  Quality of life during treatment will be measured using FACT questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: G D Murphy, MD, Principal Investigator — Situs Cancer Research Center; J Bolt, PhD, Study Director — Situs Cancer Research Center
Locations (1):
- Situs Cancer Research Center, Rogers, Arkansas, United States

REFERENCES:
- [Background] Mikirova NA, Ichim TE, Riordan NH. Anti-angiogenic effect of high doses of ascorbic acid. J Transl Med. 2008 Sep 12;6:50. doi: 10.1186/1479-5876-6-50. PMID 18789157
- [Background] Duconge J, Miranda-Massari JR, Gonzalez MJ, Jackson JA, Warnock W, Riordan NH. Pharmacokinetics of vitamin C: insights into the oral and intravenous administration of ascorbate. P R Health Sci J. 2008 Mar;27(1):7-19. PMID 18450228
- [Background] Duconge J, Miranda-Massari JR, Gonzalez MJ, Taylor PR, Riordan HD, Riordan NH, Casciari JJ, Alliston K. Vitamin C pharmacokinetics after continuous infusion in a patient with prostate cancer. Ann Pharmacother. 2007 Jun;41(6):1082-3. doi: 10.1345/aph.1H654. Epub 2007 May 22. No abstract available. PMID 17519294
- [Background] Riordan HD, Casciari JJ, Gonzalez MJ, Riordan NH, Miranda-Massari JR, Taylor P, Jackson JA. A pilot clinical study of continuous intravenous ascorbate in terminal cancer patients. P R Health Sci J. 2005 Dec;24(4):269-76. PMID 16570523
- [Background] Du J, Martin SM, Levine M, Wagner BA, Buettner GR, Wang SH, Taghiyev AF, Du C, Knudson CM, Cullen JJ. Mechanisms of ascorbate-induced cytotoxicity in pancreatic cancer. Clin Cancer Res. 2010 Jan 15;16(2):509-20. doi: 10.1158/1078-0432.CCR-09-1713. Epub 2010 Jan 12. PMID 20068072
- [Background] Levine M, Espey MG, Chen Q. Losing and finding a way at C: new promise for pharmacologic ascorbate in cancer treatment. Free Radic Biol Med. 2009 Jul 1;47(1):27-9. doi: 10.1016/j.freeradbiomed.2009.04.001. Epub 2009 Apr 8. No abstract available. PMID 19361554
- [Background] Robitaille L, Mamer OA, Miller WH Jr, Levine M, Assouline S, Melnychuk D, Rousseau C, Hoffer LJ. Oxalic acid excretion after intravenous ascorbic acid administration. Metabolism. 2009 Feb;58(2):263-9. doi: 10.1016/j.metabol.2008.09.023. PMID 19154961
- [Background] Hoffer LJ, Levine M, Assouline S, Melnychuk D, Padayatty SJ, Rosadiuk K, Rousseau C, Robitaille L, Miller WH Jr. Phase I clinical trial of i.v. ascorbic acid in advanced malignancy. Ann Oncol. 2008 Nov;19(11):1969-74. doi: 10.1093/annonc/mdn377. Epub 2008 Jun 9. PMID 18544557
- [Background] Chen Q, Espey MG, Sun AY, Lee JH, Krishna MC, Shacter E, Choyke PL, Pooput C, Kirk KL, Buettner GR, Levine M. Ascorbate in pharmacologic concentrations selectively generates ascorbate radical and hydrogen peroxide in extracellular fluid in vivo. Proc Natl Acad Sci U S A. 2007 May 22;104(21):8749-54. doi: 10.1073/pnas.0702854104. Epub 2007 May 14. PMID 17502596
- [Background] Chen Q, Espey MG, Krishna MC, Mitchell JB, Corpe CP, Buettner GR, Shacter E, Levine M. Pharmacologic ascorbic acid concentrations selectively kill cancer cells: action as a pro-drug to deliver hydrogen peroxide to tissues. Proc Natl Acad Sci U S A. 2005 Sep 20;102(38):13604-9. doi: 10.1073/pnas.0506390102. Epub 2005 Sep 12. PMID 16157892
- [Background] Chen Q, Espey MG, Sun AY, Pooput C, Kirk KL, Krishna MC, Khosh DB, Drisko J, Levine M. Pharmacologic doses of ascorbate act as a prooxidant and decrease growth of aggressive tumor xenografts in mice. Proc Natl Acad Sci U S A. 2008 Aug 12;105(32):11105-9. doi: 10.1073/pnas.0804226105. Epub 2008 Aug 4. PMID 18678913
- [Background] Ohno S, Ohno Y, Suzuki N, Soma G, Inoue M. High-dose vitamin C (ascorbic acid) therapy in the treatment of patients with advanced cancer. Anticancer Res. 2009 Mar;29(3):809-15. PMID 19414313